CLINICAL TRIAL: NCT01736267
Title: Study of Nucleus 24 and ABI541 Auditory Brainstem Implants (ABI) in Adult Non-Neurofibromatosis Type 2 Subjects
Brief Title: Auditory Brainstem Implant (ABI) in Adult Non-Neurofibromatosis Type 2 Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by IRB
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Dr. Daniel Lee, Director of Auditory Brainstem Implant Progra, Department of Otolaryngology, Massachusetts Eye and Ear Infirmary, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEEI HSC 12-061
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Bilateral Hearing Loss for Causes Other Than Tumors
Keywords: Auditory Brainstem Implant; ABI; Nucleus 24; Deafness; Hearing loss; Non-tumor; Non-NF2; ABI541
MeSH Terms: conditions — Deafness; Hearing Loss | interventions — Ankle Brachial Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Non-NF2 ABI surgery (Experimental): All subjects will be part of a single arm involving placement of the Nucleus ABI541 Auditory Brainstem Implant (ABI) device. The Nucleus 24 was discontinued and is no longer available.
  Interventions: Device: Nucleus 24 (discontinued) and ABI541 Auditory Brainstem Implants (ABI)

INTERVENTIONS:
Device: Nucleus 24 (discontinued) and ABI541 Auditory Brainstem Implants (ABI) — Nucleus ABI541 Auditory Brainstem Implant (ABI) surgery followed by device activation, testing, and clinical assessment for five years following surgery.
  Other Names: ABI, Nucleus 24, Cochlear Americas, ABI541, Nucleus Profile

SUMMARY:
The purpose of this research study is to determine whether Auditory Brainstem Implant (ABI) can improve hearing in persons who are deaf in both ears and are not candidates for cochlear implants.

DETAILED DESCRIPTION:
The goal of this MEEI Auditory Brainstem Implant (ABI) research study is to find new ways to improve hearing in patients who are deaf and cannot receive a cochlear implant. The ABI is a surgically placed bionic implant that converts sounds into electrical signals that are directly transmitted to the cochlear nucleus, the first auditory center of the brain. For many years, ABIs have improved the hearing of patients who are deaf due to brain tumors associated with a genetic syndrome called Neurofibromatosis Type 2 (NF2). However, a number of recent studies suggest that deaf patients who do not have NF2 and are not eligible for a cochlear implant may also benefit from placement of an ABI. These preliminary studies suggest that these non-NF2 or "nontumor" patients may actually have better outcomes after ABI surgery than patients suffering from NF2. Patients who do not have NF2 and are deaf due to damage to the hearing nerves or inner ears from infection, disease or injury are not cochlear implant candidates and there are no other options to improve hearing in these cases except for the ABI. Thus, the purpose of our study is to carefully analyze whether ABI surgery improves the hearing and quality of life of non-NF2 patients based on subjective and objective measures of their hearing before and after ABI surgery. In particular, we plan to study ABI outcomes in non-NF2 patients, characterize the parameters used on their devices, and determine the safety profile of ABIs in these patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English as the primary language
* Medically and psychologically suitable
* Willing to receive/have received meningitis / pneumococcal vaccinations
* Able to comply with study requirements, including travel to the investigational site
* Cochlear or retrocochlear anomaly/pathology that interferes with transmission of auditory information from the cochleae to the brainstem, resulting in severe to profound bilateral deafness (thresholds of 90 dB or worse in both ears on pure tone audiometry ranging from 250 to 2,000 Hz and speech recognition scores ≤ 30% in both ears). All subjects will undergo bone conduction audiometry and tympanometry to confirm sensorineural hearing loss and rule out potential middle ear disorders.

  * Conditions that cannot be otherwise treated, with conventional hearing aids or cochlear implants. If CI were previously used, subjects will have had a failed response, defined as ≤ 30% speech recognition and patient perception of inadequate benefit to continue using the device.
  * Expected subjects include those with these diagnoses:

    * Bilaterally severe/completely ossified cochleae
    * Bilateral cochlear malformations leading to poor CI outcomes
    * Bilateral temporal bone fractures, where the VIIIth cranial nerves have been disrupted
    * Bilateral cochlear nerve agenesis
    * Not a CI candidate based on above listed pathology, intolerable adverse effects with CI (e.g. stimulation of the facial nerve), or Evoked Auditory Potential testing predictive of a poor response

Exclusion Criteria:

* Anomalies/pathology involving the brainstem or cortex
* Retrocochlear pathology due to NF2 or other types of cranial nerve or brainstem neoplasm
* Co-existing medical conditions that require irradiation of the brainstem or auditory cortex
* Medical or psychological conditions that serve as contraindication to surgery
* Additional handicaps that would prevent or limit participation in evaluations
* Unrealistic patient or family expectations regarding the benefits, risks, and limitations inherent to the procedure and the prosthetic device
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Lee, MD, FACS, Principal Investigator — MEEI, HMS, MGH
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

REFERENCES:
- [Background] Colletti V, Shannon RV, Carner M, Veronese S, Colletti L. Complications in auditory brainstem implant surgery in adults and children. Otol Neurotol. 2010 Jun;31(4):558-64. doi: 10.1097/MAO.0b013e3181db7055. PMID 20393378
- [Background] Sennaroglu L, Ziyal I, Atas A, Sennaroglu G, Yucel E, Sevinc S, Ekin MC, Sarac S, Atay G, Ozgen B, Ozcan OE, Belgin E, Colletti V, Turan E. Preliminary results of auditory brainstem implantation in prelingually deaf children with inner ear malformations including severe stenosis of the cochlear aperture and aplasia of the cochlear nerve. Otol Neurotol. 2009 Sep;30(6):708-15. doi: 10.1097/MAO.0b013e3181b07d41. PMID 19704357
- [Background] Choi JY, Song MH, Jeon JH, Lee WS, Chang JW. Early surgical results of auditory brainstem implantation in nontumor patients. Laryngoscope. 2011 Dec;121(12):2610-8. doi: 10.1002/lary.22137. PMID 22109761
- [Background] Colletti V, Shannon R, Carner M, Veronese S, Colletti L. Outcomes in nontumor adults fitted with the auditory brainstem implant: 10 years' experience. Otol Neurotol. 2009 Aug;30(5):614-8. doi: 10.1097/MAO.0b013e3181a864f2. PMID 19546832
- See also: Related Info — http://otosurgery.org/index.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-NF2 ABI Surgery: Placement of an Auditory Brainstem Implant (ABI) device
Period: Overall Study
Arm/Group | Non-NF2 ABI Surgery
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Non-NF2 ABI Surgery
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 40 [36 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3
Pure Tone Threshold Average (dB) [Mean (Full Range); unit: dB HL] | 120 [120 to 120]

OUTCOME MEASURES:

1. Primary Outcome: Audiologic Performance
Description: Average pure tone threshold measured 12 months post-operatively. Measured in dB HL, where a lower threshold indicates more sensitive hearing and a higher threshold indicates less sensitive hearing.
  We only included data from subjects that had auditory percept of any magnitude following ABI surgery (1/3 subjects).
Time Frame: 12 months post-operative
Population: We only included data from subjects that had auditory percept of any magnitude following ABI surgery (1/3 subjects).
Measure: Number; unit: dB HL
Arm/Group | Non-NF2 ABI Surgery
Number analyzed (Participants) | 1
dB HL | 87

ADVERSE EVENTS:
Time Frame: All reported events occurred within one year of when the participant had surgery. Participants were followed through the end of their participation in the study for safety and continue to receive routine medical monitoring for safety as part of their standard care.
Arm/Group | Non-NF2 ABI Surgery
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-NF2 ABI Surgery (N=3)
Headache, photophobia, stiff neck (General disorders) | 1 (1)
clear AD drainage (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-NF2 ABI Surgery (N=3)
CSF collection (General disorders) | 1 (1) — CSF collection with mild swelling post-surgery
non-auditory side effects (Nervous system disorders) | 1 (1) — non-auditory side effects after turning on device - "pinching" sensation in the leg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT01736267/Prot_SAP_000.pdf